CLINICAL TRIAL: NCT05586841
Title: Exploration of Dalpiciclib + Chidamide in HR+/HER2- Advanced Breast Cancer After Failure of CDK4/6 Inhibitor: a Phase Ⅰb Study
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MA-BC-II-047
Record Dates: First submitted 2022-10-17; First posted 2022-10-19 (Actual); Last update posted 2022-10-19 (Actual); Status verified 2022-10

CONDITIONS: HR+/HER2- Advanced Breast Cancer
Keywords: Dalpiciclib; Chidamide; Maximum Tolerated Dose; the failure of CDK4/6 inhibitor therapy
MeSH Terms: interventions — dalpiciclib; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib + Chidamide (Experimental): Dalpiciclib will be administered in a dose of 100 mg/d or 125 mg/d. Chidamide shall be designed in a dose of 25 mg/BIW or 20 mg/BIW
  Interventions: Drug: Dalpiciclib; Drug: Chidamide

INTERVENTIONS:
Drug: Dalpiciclib — Dalpiciclib: 100 mg/d or 125 mg/d, po., qd, administered on an empty stomach (fasting should be ensured at least 1 hour before and 1 hour after administration). The drug will be administered in a 28-day cycle, with continuously administration in the first 3 weeks (D1-21), and discontinuation in the fourth week (D22-28).
  Other Names: SHR6390
Drug: Chidamide — Chidamide: 25 mg/BIW or 20 mg/BIW, po., q2w. The interval between doses should not be less than 3 days (e.g. Monday and Thursday, Tuesday and Friday, Wednesday and Saturday, etc.), administered 30 minutes after meals

SUMMARY:
A phase 1B study to explore the maximum tolerated dose (MTD) of dalpiciclib + chidamide in HR+/HER2- advanced breast cancer after the failure of CDK4/6 inhibitor therapy

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this study and sign the informed consent form
2. Female, aged ≥ 18 years.
3. ECOG PS score: 0-2 points.
4. Expected survival ≥ 3 months.
5. Regionally recurrent or metastatic disease with histologically or cytologically confirmed ER+ and/or PR+ (≥ 10%), HER2- breast cancer that is not suitable for definitive excision or radiation therapy.
6. Previously received antitumor therapy: 1) previously received ≤1 line of chemotherapy for recurrent or metastatic breast cancer; 2) Disease recurrence and/or metastasis during or after treatment with Palbociclib or Abemaciclib or Ribociclib in the setting of (neo-)adjuvant therapy, or during treatment with palbociclib or Abemaciclib or Ribociclib in a metastatic setting or after disease progression; 3) No more than 3 lines of endocrine therapy have been previously received for recurrent or metastatic breast cancer. 4) Line number of previous chemotherapy ≤1 line
7. At least one extracranial measurable lesion as defined by RECIST v1.1;
8. The function of vital organs meets the requirements;

   * Absolute neutrophil count ≥ 1.5 × 10^9/L;
   * Platelets ≥ 90 × 10^9/L;
   * Hemoglobin ≥ 90g/L;
   * Total bilirubin (TBIL) ≤ 1.5 × ULN;
   * ALT and AST ≤ 2.5 × ULN;
   * Urea/blood urea nitrogen (BUN) and creatinine (Cr) ≤1.5×ULN;
   * Left ventricular ejection fraction (LVEF) ≥ 50%;
   * The QT correction by the Fridericia formula (QTcF) is < 470 ms. INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN.
9. Subject recovers from any AE related to previous antitumor therapy before the first administration of the study drug (Grade ≤ 1).

Exclusion Criteria:

1. Previously received treatment with histone deacetylase inhibitor (HDACi);
2. Previously received Dalpiciclib;
3. MRI or lumbar puncture confirmed leptomeningeal metastasis;
4. Central nervous system metastasis is confirmed by imaging; The following conditions will be excluded: 1) asymptomatic brain metastases without immediate radiotherapy or surgery; 2) Previously received local treatment (radiotherapy or surgery) for brain metastases, stable for at least 4 weeks, and no symptomatic treatment (including glucocorticoids, mannitol, bevacizumab, etc.) for more than 2 weeks with clinical symptoms;
5. The participants presented with visceral crisis (such as lymphangitis carcinomatosis, bone marrow replacement, leptomeningeal metastasis, diffuse liver metastasis with abnormal liver function), rapid disease progression, and that is not suitable for endocrine therapy;
6. Participants had ascites, pleural effusion and pericardial effusion with clinical symptoms at baseline, which required drainage within 4 weeks before the first medication;
7. Inability to swallow, intestinal obstruction, or other factors that affect medication administration and absorption;
8. Subjects that are diagnosed with any other malignancy within 5 years prior to the study, excluding non-melanoma skin cancer treated with radical therapy, basal or squamous cell skin cancer or carcinoma in situ of the cervix and papillary thyroid.
9. The subject has undergone major surgery or major trauma or is expected to undergo major surgery within 4 weeks before the start of treatment;
10. A known history of allergy to the drug ingredient of this protocol;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Dalpiciclib + Chidamide | 2 Years
  Bayesian optimal interval (BOIN) design method will be used in this clinical trial to determine the maximum tolerated dose (MTD).

SECONDARY OUTCOMES:
Objective response rate (ORR) of different dose groups | 2 Years
  According to recist1.1 standard, the proportion of patients whose best remission was CR or PR accounted for the total number of evaluable patients.
Safety of different dose groups (incidence of treatment-related adverse events) | AE recorded from infromed consent to 28 days after treatment completion
  The severity of adverse events shall be determined according to CTCAE v5.0. During the trial, the adverse event record form should be truthfully filled in, including the occurrence time, severity, duration, measures taken and outcome of adverse events.
PFS | 2 Years
  The time from the date of randomization to the date of first documented progression or date of death from any cause, whichever came first.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China